CLINICAL TRIAL: NCT03806790
Title: Efficacy and Safety of LEO 90100 Foam in Japanese Subjects With Psoriasis Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0053-1422
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2020-11

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEO 90100 foam (Experimental): calcipotriol hydrate 52.2 µg/g [equivalent to 50.0 µg/g calcipotriol] plus betamethasone dipropionate 0.643 mg/g
  Interventions: Drug: LEO 90100 foam
- Dovobet® ointment (Active Comparator): calcipotriol hydrate 52.2 µg/g [equivalent to 50.0 µg/g calcipotriol] plus betamethasone dipropionate 0.643 mg/g
  Interventions: Drug: Dovobet® ointment

INTERVENTIONS:
Drug: LEO 90100 foam — Once daily topical application of foam from a can to psoriasis lesions. Dose depends on size of lesion.
  Other Names: Enstilar® Foam
  Arms: LEO 90100 foam
Drug: Dovobet® ointment — Once daily topical application of ointment from a tube to psoriasis lesions. Dose depends on size of lesion.
  Arms: Dovobet® ointment

SUMMARY:
Comparison of the efficacy of LEO 90100 foam with Dovobet® ointment in the treatment of psoriasis in Japanese subjects.

DETAILED DESCRIPTION:
A phase 3, national, multi-centre, 4-week, prospective, randomised, controlled, parallel-group, open trial of LEO 90100 foam versus Dovobet® ointment (both treatments containing calcipotriol hydrate plus betamethasone dipropionate) in Japanese subjects with psoriasis vulgaris.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed and dated informed consent obtained
2. Japanese subjects
3. Aged 20 years or above
4. Clinical diagnosis of psoriasis vulgaris amenable to topical treatment of less than or equal to 30% BSA (excluding psoriasis on the face/genitals/skin folds).
5. A target psoriasis lesion of at least mild severity on the body of a minimum size of 10 cm2 and scoring at least 2 (mild) for each of the clinical signs). The lesion must not be on the scalp, face, genitals or skin folds.
6. Women of childbearing potential must have a negative pregnancy test at Day 1 and agree to use an adequate methods of birth control during the trial.
7. Able to communicate with the (sub)investigator and understand and comply with the requirements of the trial.

Key Exclusion Criteria:

1. Systemic use of biological treatments with a potential effect on psoriasis vulgaris within the specified time periods prior to randomisation (depending on treatment)
2. Systemic treatments with all therapies other than biological treatments with a potential effect on psoriasis vulgaris within 4 weeks prior to randomisation
3. PUVA therapy, UVB therapy or UVA therapy on the full body or on the target lesion within 4 weeks prior to randomisation
4. Topical treatment of psoriasis on the areas to be treated with trial medication within 2 weeks prior to randomisation
5. Topical treatment of psoriasis on the face, genitals or skin folds with vitamin D3 analogues, potent corticosteroids or immunosuppressants within 2 weeks prior to randomisation
6. Topical treatment of conditions other than psoriasis with vitamin D3 analogues, potent corticosteroids or immunosuppressants within 2 weeks prior to randomisation
7. Initiation or changes of medication that may affect psoriasis vulgaris during the trial
8. Patients with certain disorders or symptoms present on the areas to be treated with trial medication: viral lesions of the skin, infections, skin manifestations, or fragility of skin veins
9. Other inflammatory skin diseases that may confound the evaluation of psoriasis vulgaris
10. Erythrodermic, exfoliative or pustular psoriasis on the areas to be treated with trial medication
11. Planned excessive exposure of areas to be treated with trial medication to either natural or artificial sunlight during the trial.
12. Disorders of calcium metabolism
13. Severe renal insufficiency, severe hepatic disorders or severe heart disease
14. Hypersensitivity to any components of the investigational medicinal products.
15. Cushing's disease or Addison's disease
16. Subjects who have received treatment with any non-marketed drug substance within the 4 weeks prior to randomisation, or longer if for certain biological treatments
17. History of cancer within the last 5 years (except completely cured skin cancer)
18. Current participation in any other interventional clinical trial
19. Previously randomised in this trial
20. Women who are pregnant, wishing to become pregnant or are breast-feeding
21. Chronic alcohol or drug abuse within 12 months prior to screening, or any condition associated with poor compliance
22. Employees of the trial site or any other individuals directly involved with the planning or conduct of the trial, or immediate family members of such individuals

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (13):
- Japan (13):
  - Leo Pharma Investigational Site, Fukutsu, Fukuoka
  - Leo Pharma Investigational Site, Obihiro, Hokkaido
  - Leo Pharma Investigational Site, Sapporo, Hokkaido
  - Leo Pharma Investigational Site, Nonoichi, Ishikawa-ken
  - Leo Pharma Investigational Site, Kawasaki, Kanagawa
  - Leo Pharma Investigational Site, Yokohama, Kanagawa
  - Leo Pharma Investigational Site, Sendai, Miyagi
  - Leo Pharma Investigational Site, Saitama-shi, Saitama
  - Leo Pharma Investigational Site, Itabashi-ku, Tokyo
  - Leo Pharma Investigational Site, Kita-ku, Tokyo
  - Leo Pharma Investigational Site, Koto-Ku, Tokyo
  - Leo Pharma Investigational Site, Minato-Ku, Tokyo
  - Leo Pharma Investigational Site, Setagaya City, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEO 90100 Foam | Dovobet® Ointment
Started | 87 | 95
Completed | 87 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 90100 Foam | Dovobet® Ointment | Total
Number analyzed (Participants) | 87 | 95 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (13.6) | 54.8 (12.9) | 54.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 58 | 61 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 87 | 95 | 182
Region of Enrollment [Number; unit: participants]
  Japan | 87 | 95 | 182

OUTCOME MEASURES:

1. Primary Outcome: Overall Improvement Rate for the Target Lesion
Description: Overall improvement defined as 'Substantial Resolution' of Clinical Signs or at Least 'Moderately Improved' in the General Change in the Lesion.
  Substantial resolution' is defined as a clinical score for thickness and scaliness of 0 and a clinical score for redness of 1 or less in the severity of clinical signs of the target lesion. The details of the clinical scores are presented in secondary outcome measure description for 'Change in the total sign score'.
  Change in the Lesion is a 5 point scale below:
  * Markedly improved (best outcome)
  * Moderately improved
  * Slightly improved
  * Unchanged
  * Aggravated (worst outcome)
Time Frame: End of Week 4
Population: The primary endpoint was analysed for the full analysis set. Rates of subjects with the event defined by the primary endpoint, 'overall improvement rate' for the target lesion at Visit 4 (end of Week 4), were compared between treatment groups by means of Fisher's exact test. Estimated rates, odds ratio, and its 95% CI were presented, together with the p-value from Fisher's exact test.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100 Foam | Dovobet® Ointment
Number analyzed (Participants) | 87 | 95
Participants | 86 | 89
Statistical Analysis 1: Comparison: LEO 90100 Foam vs Dovobet® Ointment; Statistical analysis on the Full Analysis Set (FAS); Test type: Superiority; p = 0.120, Fisher Exact; Odds Ratio (OR) = 5.80, 95% CI 2-sided [0.68 to 49.16]

2. Secondary Outcome: Overall Improvement Rate for the Target Lesion at Weeks 1 and 2
Description: Substantial resolution of clinical signs or at least 'moderately improved' in the general change in the target lesion.
  Change in the Lesion is a 5 point scale below:
  * Markedly improved (best outcome)
  * Moderately improved
  * Slightly improved
  * Unchanged
  * Aggravated (worst outcome)
Time Frame: End of Weeks 1 and 2
Population: The secondary endpoints were analysed for the full analysis set. The number and percentage of subjects with 'overall improvement' were tabulated for Visits 2 and 3 (end of Weeks 1 and 2) and by treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100 Foam | Dovobet® Ointment
Number analyzed (Participants) | 87 | 95
Participants
  Week 1 | 61 | 46
  Week 2 | 83 | 77
Statistical Analysis 1: Comparison: LEO 90100 Foam vs Dovobet® Ointment; End of Week 1 (FAS); Test type: Superiority; p = 0.004, Fisher Exact; Odds Ratio (OR) = 2.50, 95% CI 2-sided [1.36 to 4.60]
Statistical Analysis 2: Comparison: LEO 90100 Foam vs Dovobet® Ointment; End of Week 2 (FAS); Test type: Superiority; p = 0.003, Fisher Exact; Odds Ratio (OR) = 4.85, 95% CI 2-sided [1.57 to 14.97]

3. Secondary Outcome: Change in the Total Sign Score for the Target Lesion From Week 0 to Week 4
Description: The change in the total sign score from Week 0 to Week 4; total sign score is defined as the sum of the scores from the 3 clinical signs (redness, thickness, and scaliness) assessing severity in the target lesion.
  The severity for each of the 3 clinical signs was recorded according to a 9-point scale that ranges from a score of 0 to 4 in increments of 0.5; the severities are scored from low to high with 0 = none and 4 = severe. The sum of the 3 total sign scores could range from 0 (best) to 12 (worse). The greater the negative value for the change means a better outcome.
  Negative change denotes a decrease in the score and therefore a decrease in disease severity.
Time Frame: End of Week 4
Population: The secondary endpoints were analysed for the full analysis set. For the change in the total sign score, the estimated difference between the treatment groups in the mean change (LEO 90100 foam group - Dovobet® ointment group) was calculated with 95% confidence interval. The treatment difference of the change in the total sign score at Visit 4 was estimated with an ANOVA with treatment as fixed effect.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LEO 90100 Foam | Dovobet® Ointment
Number analyzed (Participants) | 87 | 95
score on a scale | -7.09 (1.48) | -5.98 (2.03)
Statistical Analysis 1: Comparison: LEO 90100 Foam vs Dovobet® Ointment; FAS; Test type: Superiority; p < 0.001, ANOVA; Estimated difference = -1.11, 95% CI 2-sided [-1.64 to -0.59]

4. Secondary Outcome: Number of Adverse Events
Description: Number of treatment emergent adverse events (TEAEs). 14-day follow-up of TEAEs was only required if the TEAE was present at the last visit, and was of possible or probable relationship to trial medication.
Time Frame: Treatment Emergent Adverse Events were assessed from Day 1 to end of Week 4, if Treatment Emergent Adverse Events were noted, they were followed for an additional 14 days
Population: The analysis of adverse events was based on the safety analysis set.
Measure: Number; unit: participants
Arm/Group | LEO 90100 Foam | Dovobet® Ointment
Number analyzed (Participants) | 87 | 95
participants | 15 | 19

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during 4 week treatment period and up to 2 weeks after the treatment period
Arm/Group | LEO 90100 Foam | Dovobet® Ointment
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/95
Other Adverse Events (participants affected / at risk) | 15/87 | 19/95
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 Foam (N=87) | Dovobet® Ointment (N=95)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Keratitis (Eye disorders) | 1 (1) | 0
Pyrexia (General disorders) | 1 (1) | 0
Bronchitis (Infections and infestations) | 0 | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0
Furuncle (Infections and infestations) | 0 | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0
Nasopharyngitis (Infections and infestations) | 5 (5) | 5 (5)
Pharyngitis (Infections and infestations) | 1 (1) | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 | 1 (1)
Blood calcium increased (Investigations) | 1 (1) | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Hypertension (Vascular disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all phase 3 clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. If no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (2):
  • Study Protocol (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03806790/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT03806790/SAP_001.pdf